CLINICAL TRIAL: NCT07156903
Title: Qualitative Erhebung Zur Erfassung Der Bedürfnisse Von Patienten Und Deren Angehörigen während Und Nach Einer Strahlentherapie Bei Prostatakarzinomerkrankung Und Deren Einstellung Und Wünsche bezüglich Einer Prähabilitationsmaßnahme
Brief Title: Evaluation of Needs of Patients and Care-givers During and After Radiotherapy of Patients With Prostate Cancer
Acronym: PrähabPro
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Prof. Dr. Franziska Hausmann, Principle Investigator, Charite University, Berlin, Germany
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: EA4/121/25
Record Dates: First submitted 2025-08-27; First posted 2025-09-05 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-09

CONDITIONS: Prostate Cancer Patients
Keywords: Qualitative Research; Prehabilitation
MeSH Terms: interventions — Interviews as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- interviews (Experimental): Patients will be asked to participate in interviews
  Interventions: Other: Interview

INTERVENTIONS:
Other: Interview — Patients and their care-givers will be asked to participate in interviews

SUMMARY:
Exploratory qualitative survey to assess the needs of patients and their relatives during and after radiotherapy for prostate cancer and their attitudes and wishes regarding prehabilitation measures

DETAILED DESCRIPTION:
Across Germany, more than 500,000 people are newly diagnosed with cancer each year (Center for Cancer Registry Data, RKI, 2020). Prostate cancer, the most common cancer in men, affects more than 65,000 patients annually (https://www.krebsinformationsdienst.de/prostatakrebs). The gold standard for the treatment of advanced prostate cancer is radiotherapy combined with anti-hormonal therapy. If the cancer is detected earlier, surgery can be performed. Both procedures are then considered to be oncologically equivalent. Despite the most modern treatment methods and techniques, severe acute and long-term side effects still occur, which patients can experience as extremely limiting. These include, among other things, loss of libido and erectile function, the development of bladder weakness and even incontinence, and changes in bowel function (e.g., diarrhea).

Currently, patients often only begin treatments designed to mitigate these side effects during their rehabilitation, at least 4-6 weeks after therapy. However, the investigators believe that greater effects can be achieved and even the occurrence of serious side effects can be potentially prevented if treatment is initiated before or during therapy. This concept is called prehabilitation.

In order to develop a suitable prehabilitation program for prostate cancer patients undergoing curative radiation therapy (either definitive or postoperative), the investigators will conduct interviews with patients and, if possible, their immediate family members (e.g., partners) to learn more about their experiences before, during, and after the treatment. The investigators would also like to learn more about their attitudes and wishes regarding prehabilitation measures.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed Prostate Cancer with curativ intended Radiotherapy
* min. 18 years
* sufficient knowledge of German language for participation in interviews
* Capacity to consent

Exclusion Criteria:

* age <18 years

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Qualitative Evaluation of Interviews | interviews will take place once either during radiotherapy or during follow up (planned 30 participants each); Each interview is expected to last 60 minutes.
  This is an exploratory, qualitative study. The data will be coded or analyzed thematically.

CONTACTS AND LOCATIONS:
Locations (1):
- Charité Universitätsmedizin Berlin, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No